CLINICAL TRIAL: NCT06707116
Title: The Mediating Role of Health Literacy in the Relationship Between Gender Differences, Illness Identity, and Self-Efficacy Patients with Cardiac Diseases: a Structural Equation Model
Brief Title: Health Literacy As a Mediator Between Gender, Illness Identity, and Self-Efficacy
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohammed Elsayed Zaky, Principal Investigator, Cairo University
Other Study IDs: Health Literacy
Record Dates: First submitted 2024-11-24; First posted 2024-11-27 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Cardiac Diseases
Keywords: Health Literacy; Gender Differences
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study group

SUMMARY:
The goal of this observational study is to understand the role of health literacy in shaping the relationship between gender differences, illness identity, and self-efficacy in geriatric patients with cardiac diseases. The main question it aims to answer is:

Does health literacy mediate the relationship between gender, illness identity, and self-efficacy in elderly cardiac patients?

Participants with diagnosed cardiac conditions, will complete online surveys assessing their health literacy, illness identity, and self-efficacy over a one-year period. Structural Equation Modeling (SEM) will be used to analyze the relationships among these variables.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 30 years or older.
* Diagnosed with a cardiac disease (e.g., heart failure, coronary artery disease, arrhythmia).
* Able to provide informed consent.
* Sufficient health literacy to complete surveys in the study language.
* Currently under regular medical care for their cardiac condition.

Exclusion Criteria:

* Individuals with a cognitive impairment or diagnosis of dementia that could interfere with survey participation.
* Patients with co-morbid terminal illnesses that significantly impact life expectancy (e.g., advanced cancer).

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients aged 30 years and older who have been diagnosed with cardiac diseases, such as coronary artery disease, heart failure, or arrhythmias. These individuals are actively receiving regular medical care for their cardiac conditions and are living in the community or non-acute care settings.
  The population includes both male and female participants to explore gender differences in illness identity, health literacy, and self-efficacy. Participants are expected to have a baseline level of health literacy sufficient to comprehend and complete the study surveys, as the research focuses on the mediating role of health literacy.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Illness Identity Questionnaire (IIQ) | 1 month
  Description: The Illness Identity Questionnaire (IIQ) is a 25-item, self-report, paper-and-pencil questionnaire that was initially used and validated in adolescents and young adults with type 1 diabetes mellitus. Patients are asked to indicate how much they agree with 25 statements, using a 5-point Likert scale ranging from 1-5 (strongly disagree to strongly agree). The IIQ consists of a 5-item rejection scale (items 1-5); 5-item acceptance scale (items 6-10); an 8-item engulfment scale (items 11-18); and 7-item enrichment scale (items 19-25).

SECONDARY OUTCOMES:
Cardiac Self-Efficacy Scale | 1 month
  The Cardiac Self-Efficacy Scale (CSES) is a valuable tool used to assess how confident individuals with heart conditions feel about managing their illness and maintaining daily activities. This scale provides insight into two main areas of self-efficacy: the ability to control symptoms, such as chest pain or fatigue, and the capacity to maintain physical and emotional well-being despite the challenges posed by their condition.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/35739464/
- See also: Related Info — https://pmc.ncbi.nlm.nih.gov/articles/PMC10944975/